CLINICAL TRIAL: NCT01031524
Title: Randomized Double-blind Controlled Phase I/IIa Trial to Assess the Efficacy of Malaria Vaccine PfCS 102 (282-383) to Protect Against Artificial Challenge With P. Falciparum
Brief Title: Trial to Assess the Efficacy of Malaria Vaccine PfCS 102
Acronym: DG002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Radboud University Medical Center (Other)
Responsible Party: Blaise Genton, Department of Ambulatory care and Community Medicine, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09/04
Record Dates: First submitted 2009-12-09; First posted 2009-12-14 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — circumsporozoite protein (282-383), Plasmodium falciparum; mannide monooleate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vaccine (Experimental): 30 µg of PfCS102 formulated in Montanide ISA 720
  Interventions: Biological: PfCS102
- adjuvant (Placebo Comparator): Montanide ISA 720
  Interventions: Biological: Montanide ISA 720

INTERVENTIONS:
Biological: PfCS102 — Antigen of the sporozoite protein
  Arms: vaccine
Biological: Montanide ISA 720 — adjuvant alone
  Arms: adjuvant

SUMMARY:
Phase I/IIa double-blind randomized (adjuvant)-controlled trial. 16 volunteers are randomized to receive two doses of either 30 µg of PfCS102 formulated in Montanide ISA 720 (verum) or ISA 720 alone (control), 60 days apart. Two weeks after the 2nd immunization, 14 volunteers are challenged with bites of 5 infected mosquitoes using the NF54 strain of P. falciparum. The main outcome will be the length of time between artificial challenge and development of blood stage parasitaemia detected by microscopy performed twice a day.

ELIGIBILITY:
Inclusion Criteria:

* resident in or near Lausanne;
* age >18 and <45 years;
* written informed consent;
* >10/12 correct responses to the questionnaire of understanding.

Exclusion Criteria:

* history of malaria; possible exposure to malaria within the previous 6 months;
* positive serology for PfCS102by ELISA;
* history of severe reactions or allergy to mosquito bites, artemether/lumefantrine (Riamet®) or vaccines;
* pregnant or lactating female;
* any confirmed or suspected immunodeficient condition;
* seropostivity for HIV;
* chronic or active neurological, gastrointestinal, cardio-vascular or respiratory disease;
* hemoglobinopathies;
* history of >2 hospitalisations for invasive bacterial infections;
* requirement of any chronic medication;
* suspected or known current alcohol or illegal drug abuse (excluding cannabis);
* any other significant finding which, in the opinion of the investigator, would significantly increase the risk of having an adverse outcome from participating in this protocol or of dropping out of the study;
* a body mass index < 18kg/m2 or > 32 kg/m2;
* evidence of past or present psychiatric condition;
* seropositivity for HIV, hepatitis C or B (other than HBs Ab);
* 10-year risk of coronary heart disease <10%;
* any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-03; Primary Completion 2004-07 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Length of time between artificial challenge and development of blood stage parasitaemia detected by microscopy | 1month

SECONDARY OUTCOMES:
Incidence of adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD PhD, Principal Investigator — University Hospital
Locations (1):
- Department of Ambulatory Care and Community Medicine; University Hospital, Lausanne, Switzerland